CLINICAL TRIAL: NCT01500291
Title: Principal Investigator
Brief Title: A Study Survey of Stress in Anesthesia Personnel
Acronym: stress
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phongthara Vichitvejpaisal", Principal Investigator, Mahidol University
Other Study IDs: 315/2554(EC3); Si445/2011 (Other: Siriraj Institutional Review Board, Mahidol University)
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Stress; Anxiety; Depression
Keywords: anesthesia stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anesthesiologist
  Interventions: Other: 2 courseware databases.
- Nurse anesthetist
  Interventions: Other: 2 courseware databases.

INTERVENTIONS:
Other: 2 courseware databases. — All participant voluntarily response all items in the SST and SAST courseware database.
  Other Names: group A; group B

SUMMARY:
It is inevitable that nearly both anesthesiologist and nurse anesthetist take a zero tolerance approach to avoidable safety problems in the provision of anesthesia.

We would like to study the stress upon anesthesia personnel by using Suanprung Stress Test (SST) - a well-documented, psychological stress test, and Siriraj Anesthesia-related Stress Test (SAST) - a new developed open-ended opinion poll, to scrutinize the daily rounds stress and yield the solution to eradicate or alleviate those worries as well as improve both physical and mental health to handle the situation of difficulties.

DETAILED DESCRIPTION:
This is a prospective study to survey the stress upon anesthesia personnel and verify causes and risk factors to their stress. A message of persuading is conducted among the anesthesia personnel in university, municipal and private hospitals. We ask participants to voluntarily response all items in questionnaires of the SST and SAST.

We launch a communication channel with the anesthesia personnel at www.nmac.in.th and require that qualified participants register and express their intention to join this research project. Each registered participant receives an identification number and a log-in password to the website containing the SST and SAST courseware database. The program is interactive, with personal files for each participant on each test along with other details like code, password, date-month-year, test scores, and log-in periods and time.

We introduced the 20 questionnaires of the SST courseware, to the developed system via http://www.dmh.go.th/test/stress/ before performing it under the research approach via www.nmac.in.th website. The findings revealed that the system operating units were flexible to participants' interactive behavior, instruction and responsiveness. Access to the system through the website provided ready access to the information, was user-friendly, and was stable. In addition, the tools were objective, covered complete details, and were clear, with elements of the subject content in proper order.

1. SST courseware comprises of 60 questionnaires with scoring through five choices: most stressful (5), highly stressful (4), moderately stressful (3), mildly stressful (2), and no stressful (1).

   In addition, the tests underwent verification for content validity and had index of item objective congruence (IOC) determined by experts; with > 0.8 in Cronbach's alpha reliability coefficient; r > 0.27 in concurrent validity through calculation of Pearson Product moment correlation against an electromyogram biofeedback.
2. SAST courseware comprises of 6 sections with scoring through visual analog scale and allowing open-ended opinions. The questionnaires had undergone quality analysis and verification for conciseness, accuracy, and clarity, as well as content and structural validity by three doctorate educational experts with at least a decade of teaching experience. The questionnaires' IOC was 0.79. The open-ended questionnaire is composed of the following sections: (1) background data: age, gender, experience in anesthesia; (2) working data: working time, overnight job, numbers of call; (3) personal data: sleeping time; (4) patient safety issues: frequency of various situations involving unsafe actions, occurrence of operating room events; (5) attitudes toward production pressure: depression, fatigue, confusion, tension/anxiety, and anger; and (6) ratings of sources of production pressure.

We ask participants to voluntarily response all items in the SST and SAST. However, they have rights not to answer any questions that put them in an awkward position.

Target group: Providing the data approximates to 1,000 anesthesiologists and 3,000 nurse anesthetists who have formally performed patient care. Participation is voluntary, without any honorarium, their only benefit is self-awareness of stress. Whether or not they participated does not affect their careers in any way.

Target group size: Two hundred and eighty six out of 1,000 anesthesiologists and three hundred and fifty three out of 3,000 nurse anesthetists are qualified as the final study group.

Procedure: After participants log in with their codes and passwords given to them, they then study the www.nmac.in.th website at their leisure for the content of the SST and SAST designed through questionnaires. Their scores are immediately provided with the completion of a testing courseware and their individual profiles updated as well. Those feeling overwhelmed by the conditions are allowed to withdraw from the project anytime.

During this research, we are willing to answer queries about the project procedure and monitor individual participants' progress through the website while keeping confidential the data about individual participants.

Information analysis:

1. A psychologist assesses the individual stress, which expressed as mean and standard deviation. All associated factors are compared by the chi-square test. Statistical significance is defined as p < 0.05.
2. Information from an open-ended questionnaire: This information yields mean and standard deviation values along with content analysis for use in our subsequent discussion.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists and nurse anesthetists who are currently working in the operating rooms.

Exclusion Criteria:

* unwilling to join the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Two hundred and eighty six out of 1,000 anesthesiologists and three hundred and fifty three out of 3,000 nurse anesthetists are qualified as the final study group.
Sampling Method: Probability Sample
Enrollment: 639 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
scores | 2 months
  A psychologist not directly involves in participants recruitment or contact and locates at a different site performs the interpretation and assessment of the individual stress.

CONTACTS AND LOCATIONS:
Overall Officials: Phongthara Vichitvejpaisal, M.D., Ph.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand